CLINICAL TRIAL: NCT05959850
Title: AMBroxol Therapy for ALS (AMBALS) Trial: a Double-blind, Randomised, Placebo-controlled Phase 2 Clinical Trial of Ambroxol for ALS
Brief Title: A Double-blind Randomised, Placebo-controlled Clinical Trial to Test Ambroxol Treatment in ALS
Acronym: AMBALS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Florey Institute of Neuroscience and Mental Health (Other)
Collaborators: Mobius Medical Pty Ltd. (Industry); The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLO-AMB-01
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-07

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Ambroxol

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial. Participants will be randomised at a 2:1 ratio to the drug solution or placebo respectively.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Active (Experimental): Ambroxol taken 3x daily. Variation in doses as follow-up progresses. For detailed information, see Intervention Description.
  Interventions: Drug: Ambroxol
- Placebo Comparator: Control (Placebo Comparator): Glucose Placebo, taken 3x daily. Variation in doses as follow-up progresses. For detailed information, see Intervention Description.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ambroxol — Participants in the study will receive varying doses of ambroxol in solution, 3 times per day. Doses will be increased pending a safety review, up to a maximum of 1260mg/day. Blood tests will be conducted weekly to assess tolerance. Compliance will be monitored by returning used bottles. The study will last 32 weeks, including 24 weeks of drug administration and follow-up visits. After the final follow-up, there will be an end of study safety visit occurring 4 weeks later. The total time of participation will be 32 weeks. This includes a screening visit up to 4 weeks prior to Baseline, then a Baseline visit, followed by 24 weeks of follow-up (3x in clinic follow-up visits). These 24 weeks will be the drug administration period, meaning that the total duration of drug administration is 24 weeks. Following this drug administration and follow-up period, there will be an EoS safety-follow up visit that will occur 4 weeks after the final follow-up visit (28 weeks from baseline).
  Other Names: Ambroxol Hydrochloride
  Arms: Experimental: Active
Drug: Placebo — Participants randomised to the control arm will receive a placebo for the duration of the study. The placebo will look and taste like ambroxol, but will have no active ingredient. Participants will not be told which arm they have been randomised to. The placebo will primarily be a glucose solution, however it will also have flavouring (e.g. bitters) and colouring, so as to make it look and taste like ambroxol, to maintain blinding.
  Arms: Placebo Comparator: Control

SUMMARY:
Ambroxol is a simple cough medicine that is predicted to slow ALS disease progression. This study aims to investigate if ambroxol in high doses is effective in treating ALS. This study will be carried out across 5 research sites in Australia (2 NSW, 1 VIC, 1 SA and 1 TAS), where newly diagnosed ALS patients will be asked to participate. Participation will be over a 32-week period, where they will come in for a 4-week screening, 24-week treatment, and 4-week end of study safety follow-up period. The participants will receive either the placebo or drug solution that they will take three times a day, up-dosing each week until they reach the maximum dose or highest dose they can tolerate. Throughout the study their disease progression will be assessed using tests, questionnaires, and blood biomarkers.

DETAILED DESCRIPTION:
This study is a double-blind, randomised, placebo-controlled phase 2 clinical trial, to assess the safety, tolerability and efficacy of ambroxol therapy in ALS patients by using electrophysiological and functional measures to detect preservation of motor units. The study design will have participants be randomised to either ambroxol or placebo at a 2:1 ratio (ambroxol (n=34) and placebo (n=16)). Participants randomised to the active arm will receive various doses of ambroxol in solution, taken orally, three times a day. Doses will be increased pending a safety review for each participant. The doses will be 180mg per day, 260mg per day, 540mg per day, 900mg per day, and 1260 mg per day. Each week safety bloods will be performed to assess tolerance to the dose. Participants randomised to the control arm will receive a placebo for the duration of the study. Disease progression will be assessed by the following, time to event (death, need for tracheostomy, the need for gastrostomy feeding or non-invasive ventilation support (≥12 hours a day in a 24-hour period), or ≥6-point progression (ALS functional rating score-revised).

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study related assessments are performed and must be able to understand purpose of the study, including any possible risks and adverse events.
2. ALS as diagnosed according to the recently proposed Gold Coast diagnostic criteria.
3. First symptom of ALS less than or equal to 18 months prior to screening. The qualifying first symptoms of ALS are limited to manifestations of weakness in extremity, bulbar, or respiratory muscles. Cramps, fasciculations, or fatigue should not be taken in isolation as a first symptom of ALS.
4. Forced vital capacity (FVC) greater than or equal to 60% of predicted value as adjusted for gender, height and age at the Screening Visit.
5. Male or female patients aged 18 years or greater (inclusive) and less than 85 years at the time of ALS diagnosis.
6. Able to swallow liquid.
7. Able to perform reproducible pulmonary function tests
8. Female patients must be post-menopausal or sterilized or must not be breastfeeding, have no intention to become pregnant during the study, and use acceptable methods of contraception or abstain from intercourse.
9. Male patients who have not had a vasectomy and confirmed zero sperm count must agree after receiving the first dose of study drug either to use acceptable methods of contraception or abstain from intercourse.
10. If on riluzole, stable dosing for 30-days prior to screening.
11. Pre-study ALSFRS-R progression between disease onset and screening of greater than or equal to 0.5 points/month (calculated by ALSFRS-R total score decline from 48 divided by the months since onset of ALS symptoms).

Exclusion Criteria:

1. Use of non-invasive ventilation (NIV) support for ALS only or gastrostomy tube at time of screening.
2. Exposure to investigational drug within 12-weeks prior to screening.
3. At screening of any medically significant cardiac, pulmonary, GI, musculoskeletal, or psychiatric illness that might interfere with the patient's ability to comply with study procedures or that might confound the interpretation of clinical safety or data.
4. Patient with a history of significant other major medical conditions based on the Investigator's judgment.
5. Based on the investigator's judgment, patients who may have difficulty complying with the protocol and/or any study procedures.
6. Any person who is an employee or an Investigator or Sponsor, or an immediate relative of an Investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Time to event | Time to event for a maximum of 24 weeks from baseline
  Time to event (death, need for tracheostomy, the need for gastrostomy feeding or non-invasive ventilation (NIV) support (greater than or equal to 12 hours a day in a 24-hour period), or greater than or equal to 6-point progression on the Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS)) This will be measured by patient medical records, and the completion of the ALSFRS by investigators.

SECONDARY OUTCOMES:
ALS functional rating score-revised (ALSFRS-R) | 24 weeks from Baseline
  Change in ALSFRS-R Score
Motor unit number estimation (MUNIX) | 24 weeks from Baseline
  Change in MUNIX values
Split Hand Index (SI) | 24 weeks from Baseline
  Change in SI value
Neurophysiology Index (NPI) | 24 weeks from Baseline
  Change in NPI Value
Kings staging system | 24 weeks from Baseline
  Change in Kings stage
Muscle strength assessment as measured by the Medical Research Council (MRC) Scale for Muscle Strength | 24 weeks from Baseline
  Change in Muscle strength, where Grade 0 is no visible contraction and Grade 5 is Normal
Respiratory function (FVC) as measure by a Spirometer | 24 weeks from Baseline
  Change in FVC
Survival | 24 weeks from Baseline
  Overall survival rate
Serum NFL levels | 24 weeks from Baseline
  Change in Serum NFL Levels
Assessment of Quality of Life (AQoL) | 24 weeks from Baseline
  Change in AQoL score

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Turner, Study Chair — The Florey Institute of Neuroscience and Mental Health; Steve Vucic, Principal Investigator — Concord Repatriation General Hospital; Matthew Kiernan, Principal Investigator — Brain and Mind Centre (The University of Sydney); Susan Mathers, Principal Investigator — Calvary Health Care Bethlehem; David Schultz, Principal Investigator — Flinders Medical Centre; Lauren Giles, Principal Investigator — Launceston General Hospital
Locations (5):
- Australia (5):
  - Brain and Mind Centre, Sydney, New South Wales
  - Concord Repatriation General Hospital, Sydney, New South Wales
  - Flinders Medical Centre, Adelaide, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Calvary Health Care Bethlehem, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
No plan to have individual participant data available to other researchers